CLINICAL TRIAL: NCT07220239
Title: Menstrual Cup-based Endometrial Collection as an Alternative to Endometrial Biopsy in Lynch Syndrome Patients
Brief Title: Menstrual Cup for Early Endometrial Cancer Detection in Lynch Syndrome
Acronym: SCREEN-CUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica D. St. Laurent, MD (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Jessica D. St. Laurent, MD, Director, Gynecologic Oncology Laboratory, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25-416
Record Dates: First submitted 2025-08-11; First posted 2025-10-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer; Lynch Syndrome; Screening; Early Detection of Cancer
Keywords: Endometrial Cancer; Lynch Syndrome; Screening; Early detection; Organoids
MeSH Terms: conditions — Endometrial Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Intervention Model Description: Pre-Pilot study: one study arm with healthy women Main Pilot study: one study arm with Lynch syndrome carriers
Masking Description: Only one part of the outcome assessor will be masked: the pathologist evaluating the EMB specimen and menstrual cup-collected specimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pilot study arm (Other): Single arm study: Intervention includes use of a mentrual cup to collect menstrual fluid
  Interventions: Device: Menstrual cup use

INTERVENTIONS:
Device: Menstrual cup use — Menstrual cup use in menstruating women to collect menstrual fluid with the aim to 1) compare the histology to endometrial biopsy samples from the same patient, to 2) investigate the feasibility and clinical utiliy of a menstrual cup use as a screening method for endometrial cancer and to 3) generate organoids from the menstrual cup samples

SUMMARY:
Study Goal:

This pilot study wants to find out if using a menstrual cup can be a good, non-invasive way to collect samples from the lining of the uterus (called the endometrium) to help screen for endometrial cancer. This is especially important for women who have a higher chance of getting this cancer, such as those with a genetic condition called Lynch syndrome.

Main Questions the Study Will Answer:

1. Can a menstrual cup collect enough uterine lining (endometrial tissue) for doctors to examine under a microscope?
2. Are the samples from the menstrual cup as useful for diagnosis as samples taken using the usual method (called an endometrial biopsy or EMB)?
3. Is using a menstrual cup at home easy, effective, and comfortable for participants?
4. Can scientists grow small lab models of the uterus (called organoids) from the menstrual cup samples and from biopsy samples?

What Will Happen in the Study:

* Participants will use a menstrual cup at home to collect menstrual blood.
* They will also have a standard endometrial biopsy done by a healthcare provider.
* After both collections, participants will fill out a short survey about how comfortable and easy it was to use the menstrual cup.

What the Study Will Measure:

* Feasibility: How well participants are able to use the menstrual cup and send in the sample.
* Sample Quality: Whether the menstrual cup collects enough good-quality tissue for testing, and how it compares to biopsy samples.
* Participant Experience: How women feel about using the menstrual cup, based on the survey.
* Lab Testing: Whether researchers can successfully grow endometrial organoids from both types of samples.

Why This Study Matters: If this method works, it could offer a gentler, more convenient way for women to get checked for endometrial cancer-especially those who need regular screening. It could also make it easier to collect samples for research and improve early detection of cancer.

DETAILED DESCRIPTION:
Menstrual Cup for Early Endometrial Cancer Detection in Lynch Syndrome (SCREEN-CUP) The study entails two parts that will be conducted one after each other.

1. Pre-pilot study Pre-pilot study including 5 menstruating females who will provide a one-time menstrual cup-based endometrial collection for the generation of organoids and for a pathological evaluation of endometrial specimen from menstrual fluid.

   After optimizing the study protocol in the pre-pilot study period, the main study will be conducted.
2. Main pilot study Prospective feasibility study including 20 female LS carriers undergoing annual endometrial biopsy for endometrial cancer surveillance or suspected endometrial pathology will provide a one-time menstrual cup-based endometrial collection and endometrial biopsy specimen. One study aim is to evaluate the comparability and quality of the menstrual cup-based endometrial collection with the EMB sample from the same patient. For the second study aim, endometrial sample collected with the menstrual cup and EMB will be used and compared for organoid generation. Patient satisfaction and feasibility will be monitored through patient and provider questionnaires.

ELIGIBILITY:
Pre-pilot study

Inclusion criteria:

* Individuals over the age of 18
* Menstruating

Exclusion criteria:

* Levonorgestrel IUD in situ or removed within the last 30 days prior to sample collection
* Patients with prior endometrial ablation
* Prior history of endometrial cancer or endometrial intraepithelial neoplasia
* History of germline pathologic germline variant in MLH1, MSH2, MSH6, PMS2, or EPCAM
* Known allergy against menstrual cup material (silicone)

Main Study Inclusion criteria

* LS carrier with a pathogenic or likely pathogenic germline variant in MLH1, MSH2, MSH6, PMS2, or EPCAM
* Individuals over the age of 18
* Planned screening EMB
* Menstruating
* Ability to give consent

Exclusion criteria:

* Current pregnancy
* Levonorgestrel IUD in situ or removed within the last 30 days prior to sample collection
* Patients with prior endometrial ablation
* Prior history of endometrial cancer
* Known allergy against menstrual cup material (silicone)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of samples considered adequate for pathologic evaluation | Postprocedural (7-14 days after study visit #2)
  A pathologist will evaluate the menstrual cup-based sample and record its adequacy for pathological evaluation using a questionnaire with binary responses.

SECONDARY OUTCOMES:
Overall participant satisfaction with menstrual cup collection for endometrial screening. | Periprocedural (on day of study visit #2)
  Participants self-report to questions on overall participant satisfaction with menstrual cup collection for endometrial screening with 5 answer possiblities ranging from "very satisfied" to "very dissatisfied".
Successful endometrial organoid generation from menstrual cup sample | Postprocedural (5-7 days after study visit #2)
  Successful organoid generation from menstrual cup sampleswill be assessed by viability assays after 5 days of culture and immunofluorescence imaging to compare cell composition.
Successful endometrial organoid generation from endometrial biopsy sample (EMB). | Postproceduaral (5-7 days after study visit #2)
  Successful organoid generation from EMB samples will be assessed by viability assays after 5 days of culture and immunofluorescence imaging to compare cell composition.
Provider satisfaction of menstrual cup collection for endometrial cancer screening within this study setting | Through study completion, an average of 1 year.
  Provider self-report on question regarding satisfaction of menstrual cup collection for endometrial cancer screening within this study setting with 5 answer possiblities ranging from "very satisfied" to "very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D St. Laurent, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a data use agreement. The protocol and statistical analysis plan will be made available to on clinicaltrials.gov only as required by federal regulations or as a condition of awards and agreements supporting research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months after publication of the primary results, for a period of up to 3 years.
Access Criteria: Researchers must submit a methodologically sound proposal and demonstrate an IRB-approved protocol. Requests maybe directed to the sponsor investigator or designee. A formal data use agreement will be required prior to access.
URL: https://www.stlaurentlab.org/

REFERENCES:
- [Background] Cindrova-Davies T, Zhao X, Elder K, Jones CJP, Moffett A, Burton GJ, Turco MY. Menstrual flow as a non-invasive source of endometrial organoids. Commun Biol. 2021 Jun 17;4(1):651. doi: 10.1038/s42003-021-02194-y. PMID 34140633
- [Background] Jenkins RW, Aref AR, Lizotte PH, Ivanova E, Stinson S, Zhou CW, Bowden M, Deng J, Liu H, Miao D, He MX, Walker W, Zhang G, Tian T, Cheng C, Wei Z, Palakurthi S, Bittinger M, Vitzthum H, Kim JW, Merlino A, Quinn M, Venkataramani C, Kaplan JA, Portell A, Gokhale PC, Phillips B, Smart A, Rotem A, Jones RE, Keogh L, Anguiano M, Stapleton L, Jia Z, Barzily-Rokni M, Canadas I, Thai TC, Hammond MR, Vlahos R, Wang ES, Zhang H, Li S, Hanna GJ, Huang W, Hoang MP, Piris A, Eliane JP, Stemmer-Rachamimov AO, Cameron L, Su MJ, Shah P, Izar B, Thakuria M, LeBoeuf NR, Rabinowits G, Gunda V, Parangi S, Cleary JM, Miller BC, Kitajima S, Thummalapalli R, Miao B, Barbie TU, Sivathanu V, Wong J, Richards WG, Bueno R, Yoon CH, Miret J, Herlyn M, Garraway LA, Van Allen EM, Freeman GJ, Kirschmeier PT, Lorch JH, Ott PA, Hodi FS, Flaherty KT, Kamm RD, Boland GM, Wong KK, Dornan D, Paweletz CP, Barbie DA. Ex Vivo Profiling of PD-1 Blockade Using Organotypic Tumor Spheroids. Cancer Discov. 2018 Feb;8(2):196-215. doi: 10.1158/2159-8290.CD-17-0833. Epub 2017 Nov 3. PMID 29101162
- [Background] Hewitt SC, Dickson MJ, Edwards N, Hampton K, Garantziotis S, DeMayo FJ. From cup to dish: how to make and use endometrial organoid and stromal cultures derived from menstrual fluid. Front Endocrinol (Lausanne). 2023 Sep 21;14:1220622. doi: 10.3389/fendo.2023.1220622. eCollection 2023. PMID 37810883